CLINICAL TRIAL: NCT05766761
Title: Designing a Hybrid Intervention Strategy to Reduce Alcohol Exposed Pregnancies
Brief Title: Reducing Alcohol Exposed Pregnancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); Health Resources in Action, Inc. (Other); Purdue University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U01AA030187-01 (NIH)
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Drinking
Keywords: alcohol drinking in pregnancy; alcohol-exposed pregnancies; alcohol-related adverse birth outcomes
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: Eligible women are randomized to either (1) the intervention condition, the usual prenatal plus the alcohol intervention, or (2) the comparison condition, usual prenatal care only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention condition, the usual prenatal care plus the alcohol intervention (Experimental): The alcohol intervention consists of (1) a self-paced computer-delivered component to enhance knowledge, norms, and motivation for alcohol reduction and (2) a nurse-delivered component to reinforce the computer-delivered content and address women's questions.
  Interventions: Behavioral: Intervention condition, the usual prenatal care plus the alcohol intervention
- Comparison condition, usual prenatal care only (No Intervention): Prenatal usual care involves clinicians assessing alcohol use and counseling women on alcohol-related risks.

INTERVENTIONS:
Behavioral: Intervention condition, the usual prenatal care plus the alcohol intervention — The intervention is theory-driven, based on Motivational Enhancement Theory (MET), and uses motivational strategies to promote alcohol reduction.
  Arms: Intervention condition, the usual prenatal care plus the alcohol intervention

SUMMARY:
The goal of this clinical trial is to compare an active intervention versus a standard of care control in reducing alcohol use among pregnant women. The main questions it aims to answer are whether a motivational intervention can:

1. increase the proportion of women detected with a laboratory-confirmed negative phosphatidylethanol (PEth) test during pregnancy, and
2. reduce the proportion of adverse birth outcomes among infants. Participants will be offered (1) a self-paced computer-delivered alcohol reduction intervention to enhance knowledge, norms, and motivation for alcohol reduction and (2) a nurse-delivered component to reinforce the computer-delivered content and address women's questions. Both components are theory-driven, based on Motivational Enhancement Theory (MET), and use motivational strategies to promote alcohol reduction.

DETAILED DESCRIPTION:
Prenatal alcohol exposure (PAE) increases the risk for Fetal Alcohol Spectrum Disorders (FASD). To address this health threat, researchers at New York University (NYU), the University of Texas Health Science Center-Houston, Purdue University, Health Resources in Action and the Collaborative Initiative on Fetal Alcohol Spectrum Disorders (CIFASD) will develop, implement, and evaluate an alcohol intervention for women in prenatal care. This study is a randomized controlled trial (N=600) to assess the efficacy of an alcohol intervention, relative to usual prenatal care only, in reducing (1) women's alcohol use and 2) poor infant birth outcomes. We will recruit women at their first prenatal care visit. Eligible women complete a baseline assessment by a research nurse consisting of an Audio Computer-Assisted Self Interview (ACASI) and collection of bloodspots for phosphatidylethanol (PEth) analysis to assess alcohol consumption biologically. Subsequently, women are randomized to either (1) the intervention condition, the usual prenatal plus the alcohol intervention, or (2) the comparison condition, usual prenatal care only. Prenatal usual care involves clinicians assessing alcohol use and counseling women on alcohol-related risks. The alcohol intervention consists of (1) a self-paced computer-delivered component to enhance knowledge, norms, and motivation for alcohol reduction and (2) a nurse-delivered component to reinforce the computer-delivered content and address women's questions. Both components are theory-driven, based on Motivational Enhancement Theory (MET), and use motivational strategies to promote alcohol reduction. The alcohol intervention is developed with guidance from multiple sources, including (1) the project's Women's Advisory Board; recruited from the proposed recruitment clinics who self-report alcohol use during pregnancy, and (2) project investigators and consultants with extensive experience and expertise in research and trial design, and developing and implementing Screening, brief intervention and referral to treatment (SBIRTs) for reducing alcohol use and other drugs among women, including pregnant women. The alcohol intervention is delivered on three occasions: (1) following the baseline and the 2nd- and 3rd-trimester assessments. Women randomized to receive usual prenatal care only complete assessments on the same schedule as women in the intervention condition. We will use generalized estimating equation models and an intent-to-treat analysis to evaluate the efficacy of the intervention condition relative to the usual prenatal care condition in (1) increasing the proportion of women detected with a laboratory-confirmed negative PEth test during pregnancy and (2) reducing the proportion of adverse birth outcomes among infants. The proposed research is scientifically and clinically significant. If demonstrated effective, the intervention may represent a scalable alcohol reduction strategy suitable for prenatal clinical care in other maternity hospitals and clinical sites to reduce prenatal alcohol exposure and adverse birth outcomes. If successful, this would be the first prevention intervention for CIFASD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Gestational age is 28 weeks or less
* Recent alcohol use as assessed by self-report of alcohol use in the previous 30 days

Exclusion Criteria:

* Under 18 years of age
* Not pregnant or gestational age over 28 weeks
* No recent alcohol use as assessed by self-report

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Can get pregnant
Enrollment: 600 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Negative PEth among women | Through study completion, on average 6 months post-enrollment
  Proportion of women detected with a laboratory-confirmed negative PEth test during pregnancy

SECONDARY OUTCOMES:
Pre-term births | At birth
  Proportion of infants whose gestational age is <37 weeks
Low birth weight | At birth
  Proportion of infants who weighed less than 2500 grams at birth

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DiClemente, PhD, Principal Investigator — New York University
Locations (1):
- The University of Texas Health Science Center, Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IDP will be shared to other researchers as part of the CIFASD data sharing protocol
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available after the study completion for a period of 5 years
Access Criteria: Will be available via the CIFASD data repository

REFERENCES:
- [Derived] Capasso A, Stotts AL, Xu MA, Manuel BD, Zelaya S, Casillas SJ, Villarreal YR, Dorow A, Brown JL, Xu S, Concheiro-Guisan M, Fonseca Pego AM, Wingood GM, Beegle SAP, DiClemente RJ; Collaborative Initiative on Fetal Alcohol Spectrum Disorders (CIFASD). Safe start, a hybrid intervention to reduce alcohol exposed pregnancies: protocol for a randomized controlled trial. BMC Public Health. 2026 Jan 10;26(1):506. doi: 10.1186/s12889-025-26044-2. PMID 41520132